CLINICAL TRIAL: NCT04053192
Title: Contemporary Use of Percutaneous Balloon Aortic Valvuloplasty and Evaluation of Its Success in Different Hemodynamic Entities of Severe Aortic Valve Stenosis
Brief Title: Evaluation of BAV in Different Hemodynamic Entities of Severe AS
Acronym: BAV
Status: Completed | Type: Observational
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Other Study IDs: 19-003 BAV
Record Dates: First submitted 2019-08-07; First posted 2019-08-12 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Aortic Valve Stenosis
Keywords: Balloon Aortic Valvuloplasty; Severe Aortic Valve Stenosis; Surgical aortic valve replacement (SAVR)
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- High-Gradient Aortic Stenosis (HG-AS): (Pmean >40mmHg, AVA <1cm^2, Vmax >4m/s)
  Interventions: Procedure: BAV; Procedure: BAV + TAVR; Procedure: SAVR
- Low-Flow-Low-Gradient Aortic Stenosis (LF-LG): (Pmean <40mmHg, AVA <1cm^2, Vmax <4m/s, EF <50%)
  Interventions: Procedure: BAV; Procedure: BAV + TAVR; Procedure: SAVR
- Paradoxe Low-Flow Low Gradient Aortic Stenosis (pLF-LG AS): Pmean <40mmHg, AVA <1cm^2, Vmax < 4m/s, EF >50%)
  Interventions: Procedure: BAV; Procedure: BAV + TAVR; Procedure: SAVR

INTERVENTIONS:
Procedure: BAV — BAV
Procedure: BAV + TAVR — BAV + TAVR
Procedure: SAVR — Surgical aortic valve replacement (SAVR)

SUMMARY:
The purpose of this retrospective, observational study is to compare the profit of BAV and TAVI in different subtypes of serve aortic stenosis.

DETAILED DESCRIPTION:
The Balloon Aortic Valvuloplasty (BAV) is a catheter-based intervention, which can be used for dilatation of serve aortic stenosis. With this minimally invasive intervention an increase of the aortic valve area (AVA) and cardiac ejection fraction (EF), decrease of transvalvular gradients and ultimately a symptom relief should be achieved. The required effect is temporary and a definitive treatment should be aspired in suitable patients. Therefor Transcatheter Aortic Valve Replacement (TAVR) is available.

Following the guidelines of the European Society of Cardiology for the management of valvular heart disease from 2017, the aortic stenosis can be divided into different subtypes by using haemodynamic parameters: High-gradient AS (HG-AS), Low-Flow-Low-Gradient AS (LFLG-AS) and paradoxical Low-Flow-Low-Gradient (pLFLG-AS). Patients with LFLG-AS are suspected to have a poorer prognosis when treated curative as well as when treated palliative medicamentous, because these patients show coronary and myocardial restrictions more frequently in addition to the valvular disease.

The aim of the study is to compare safety and effectiveness of balloon aortic valvuloplasty as a bridging therapy and transcatheter aortic valve replacement as a definitive treatment in HG-AS, LFLG-AS and pLFLG-AS patients to verify whether the subtypes of aortic stenosis profit equally from these interventions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Severe Aortic Stenosos who underwent BAV

Exclusion Criteria:

* insufficient echocardiographic parameters before BAV

Ages: 50 Years to 97 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in the heart failure program of the University of Duesseldorf
Sampling Method: Non-Probability Sample
Enrollment: 166 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
All-cause Mortality | 1-Year post BAV
Post-Procedure Hemodynamic Changes | 24 - 72 h after procedure
  dPmean, dPmax, AVA, Vmax, EF; Evaluation by using the first echocardiographic parameters after BAV / TAVR

SECONDARY OUTCOMES:
Number of patients with myocardial infarction | 30 days after intervention
  Evaluation by using the VARC-2 definition
Number of patients with stroke | 30 days after intervention
  Evaluation by using the VARC-2 definition
Number of patients with bleeding complications | 30 days after intervention
  Evaluation by using the VARC-2 definition
Number of patients with acute kidney injury | 30 days after intervention
  Evaluation by using the VARC-2 definition
Number of patients with vascular complications | 30 days after intervention
  Evaluation by using the VARC-2 definition

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Zeus, MD, Principal Investigator — Div. of Heinrich-Heine-University, Div. of Cardiology, Pulmonary Disease and Vascular Medicine
Locations (1):
- Division of Cardiology, Pulmonary Disease and Vascular Medicine, Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: Undecided